CLINICAL TRIAL: NCT06738693
Title: External Fixation Versus Volar Locking Plate for Unstable Intraarticular Distal Radius Fractures: a Prospective Comparative Study of the Functional Outcomes
Brief Title: External Fixation Vs. Volar Plate for Distal Radius Fractures: Functional Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Sabir Kumar Khadka, Junior Resident, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRC/1656/019
Record Dates: First submitted 2024-12-05; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Radius Fractures
MeSH Terms: conditions — Radius Fractures | interventions — External Fixators; Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- External Fixation (Experimental): Patients in this arm will undergo external fixation for unstable intra-articular distal radius fractures. The procedure involves the placement of an external fixator to stabilize the fracture, followed by postoperative care including pin tract cleaning and removal of the fixator after radiological confirmation of bone healing (6-8 weeks). Functional outcomes, fracture union, and complications will be assessed at regular intervals.
  Interventions: Procedure: External Fixation
- Volar Locking Plate (Experimental): Patients in this arm will undergo open reduction and internal fixation (ORIF) using a volar locking plate for unstable intra-articular distal radius fractures. This method provides stable fixation, allowing early mobilization. Postoperative outcomes, including functional scores, union rates, and complications, will be evaluated at follow-up visits.
  Interventions: Procedure: Open Reduction and Internal Fixation (ORIF) with Volar Locking Plate

INTERVENTIONS:
Procedure: External Fixation — External fixation involves the stabilization of unstable intra-articular distal radius fractures using an external fixator. The procedure is performed under anesthesia, with fixator pins placed percutaneously into the proximal and distal fragments of the radius. Postoperative care includes regular cleaning of pin tracts, early mobilization exercises for adjacent joints, and fixator removal upon radiological confirmation of fracture healing, typically between 6 to 8 weeks post-surgery.
  Arms: External Fixation
Procedure: Open Reduction and Internal Fixation (ORIF) with Volar Locking Plate — ORIF using a volar locking plate is performed to anatomically reduce and stabilize unstable intra-articular distal radius fractures. The procedure is conducted under anesthesia, involving an open approach through the volar aspect of the wrist. The volar locking plate is secured with screws to provide rigid fixation, enabling early mobilization. Postoperative follow-up includes evaluation of functional outcomes, union rates, and potential complications.
  Arms: Volar Locking Plate

SUMMARY:
The goal of this prospective comparative clinical trial is to evaluate the effectiveness of external fixation versus volar locking plates in the management of unstable intra-articular distal radius fractures in adults over 18 years old. The main questions it aims to answer are:

Does the use of a volar locking plate result in better functional outcomes, as measured by the Green and O'Brien scoring system modified by Cooney, compared to external fixation? What are the differences in intraoperative and postoperative parameters, including complications, between the two methods? Researchers will compare outcomes in two groups: one receiving external fixation and the other undergoing open reduction and internal fixation with volar locking plates.

Participants will:

Undergo surgical intervention (external fixation or ORIF with volar plates) performed by experienced orthopedic surgeons.

Follow a postoperative rehabilitation plan, including active and passive range of motion exercises.

Attend follow-ups at 6, 12, and 24 weeks to assess pain, range of motion, fracture union, and complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Diagnosed with recent (<1 week) intra-articular distal end radius fractures.
* Willing and able to provide informed consent.

Exclusion Criteria:

* Open fractures classified as Gustilo grade II or higher.
* Fracture avulsion or dislocation.
* Vascular injury associated with the fracture.
* Extra-articular fractures of the distal radius.
* Preexisting joint or carpal bone disease affecting rehabilitation.
* Patients unwilling to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2020-09-12 (Actual); Study Completion 2020-11-14 (Actual)

PRIMARY OUTCOMES:
Functional Outcomes Assessed by the Green and O'Brien Scoring System Modified by Cooney | 24 weeks post-surgery
  The primary outcome will be the functional outcome of the wrist assessed using the Green and O'Brien scoring system modified by Cooney. This scoring system evaluates four components: pain, function, range of motion, and grip strength, each weighted appropriately to provide a composite score. Scores will be compared between the external fixation and volar plating groups to determine the superiority of either intervention in restoring wrist function.

CONTACTS AND LOCATIONS:
Locations (1):
- BPKIHS, Dharān, Koshi, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) will be shared with other researchers upon reasonable request.